CLINICAL TRIAL: NCT03670095
Title: Interventional, Randomized, Single-dose, Open-label, Crossover, Bioequivalence Study in Healthy Subjects to Compare Two Pharmaceutical Formulations of Memantine (Ebixa®) in Fasted and Fed Conditions
Brief Title: Study in Healthy Subjects to Compare Two Tablet Formulations of Memantine (Ebixa®) in Fasted and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17773A
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactose-free memantine tablet (Experimental): (treatment A - test) - 10 mg; orally as a single dose in fed and fasted state
  Interventions: Drug: Lactose-free memantine
- Lactose-containing memantine tablet (Ebixa®) (Experimental): (treatment B - reference) - 10 mg, orally as a single dose in fed and fasted state
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Lactose-free memantine — Lactose-free memantine tablet, 10 mg; orally as a single dose
  Arms: Lactose-free memantine tablet
Drug: Memantine — Lactose-containing memantine tablet, 10 mg, orally as a single dose
  Other Names: Ebixa®
  Arms: Lactose-containing memantine tablet (Ebixa®)

SUMMARY:
The purpose of this study is to investigate the release of memantine into the bloodstream of two different formulations: one formulation containing lactose and one without lactose.

DETAILED DESCRIPTION:
The study consists of two cohorts: A1 and A2.

Subjects in Cohort A1 will be administered the investigational medicinal product (IMP) in a fasted state and subjects in Cohort A2 will be administered the IMP in a fed state.

Each subject will change cohort during study participation, so that dosing will be done over two periods: either first fed and then fasted, or first fasted and then fed. The two periods will be separated by a period of 28 days (+7 days) where no investigational medicinal product is given.

All subjects will be confined to the clinic from one day prior to dosing until Day 4 (72 hours post-dose) in each dosing period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women ≥18 years of age with a body mass index (BMI) ≥18.5 and ≤28 kg/m2.
* Women must be non-pregnant and non-lactating.

Exclusion Criteria:

- The subject has any concurrent disorder that may affect the particular target or absorption, distribution, or elimination of the IMP.

Other in- and exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
AUC0-72h in fed state for test and reference treatment | From zero to 72 hours post dose
  Area under the memantine plasma concentration-time curve
AUC0-72h in fasted state for test and reference treatment | From zero to 72 hours post dose
  Area under the memantine plasma concentration-time curve
Cmax of memantine in fed state for test and reference treatment | From zero to 72 hours post dose
  Maximum observed plasma concentration of memantine
Cmax of memantine in fasted state for test and reference treatment | From zero to 72 hours post dose
  Maximum observed plasma concentration of memantine

SECONDARY OUTCOMES:
tmax in fed state for test and reference treatment | From zero to 72 hours post dose
  Nominal time corresponding to the occurrence of Cmax
tmax in fasted state for test and reference treatment | From zero to 72 hours post dose
  Nominal time corresponding to the occurrence of Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Shuguang Hospital, Shanghai TCM University, Shanghai, China